CLINICAL TRIAL: NCT07199283
Title: The PEPP Trial: A Postpartum Bundle Intervention to Improve Cardiometabolic Health in Women After a First Pregnancy Affected by Preeclampsia - a Multi-centre Randomised Controlled Trial
Brief Title: The PreEclampsia Postpartum Prevention Trial
Acronym: PEPP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Kari Johansson, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2024-03584-01
Record Dates: First submitted 2025-08-14; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Preeclampsia; Postpartum Period; Hypertension; Cardiovascular Diseases; Overweight; Obesity
Keywords: Preeclampsia; Postpartum prevention; Prevention cardiometabolic disease; Hypertension; Postpartum weight loss
MeSH Terms: conditions — Pre-Eclampsia; Hypertension; Cardiovascular Diseases; Overweight; Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): Standard care
- Bundle Intervention (Experimental): Bundle Intervention
  Interventions: Other: Bundle Intervention

INTERVENTIONS:
Other: Bundle Intervention — Bundle intervention
  Arms: Bundle Intervention

SUMMARY:
The goal of this clinical trial is to learn if a postpartum bundle intervention can improve cardiometabolic health and lifestyle-related factors in women who have had preeclampsia during their first pregnancy. The main questions it aims to answer are:

* Does the 9-month intervention reduce systolic and diastolic blood pressure?
* Does the intervention promote postpartum weight loss?
* Does the intervention affect weight and blood pressure depending on early pregnancy BMI? Researchers will compare the bundle intervention to standard care to see if the intervention improves cardiometabolic health and lifestyle outcomes.

All participants will attend clinical visits for outcome assessments.

Participants in the intervention group will:

* Receive online targeted screening and group meetings with study personnel
* Use the trial-specific PEPP app to access self-monitoring tools for blood pressure and weight, lifestyle modification, and health education
* Follow the intervention in two phases: starting after inclusion (≈8 weeks postpartum) with a Light phase (baseline-3 months) and progressing to an Intensive phase (3-9 months)

DETAILED DESCRIPTION:
PURPOSE AND AIMS:

The overall aim of this 9-month multicentre, two-arm, single-blind, parallel-group RCT across several regions in Sweden is to improve cardiometabolic health in women after a first pregnancy complicated by preeclampsia, through a bundle intervention of combined evidence-based components delivered primarily via a trial-specific mobile health (mHealth) app.

The primary aim of the 9-months PEPP (PreEclampsia Postpartum Prevention) randomized controlled trial (RCT) is to evaluate if a bundle intervention is more effective than standard postpartum care in reducing systolic and diastolic blood pressure levels among first-time mothers with a recent diagnosis of preeclampsia.

Secondary aims are to evaluate whether the bundle intervention, compared to standard care, leads to greater postpartum weight loss (i.e. reduction of pregnancy-related weight gain), and greater reduction in blood pressure and weight when stratified by early pregnancy body mass index (BMI) <25/≥25 kg/m2.

Exploratory aims are to evaluate if the intervention improves the identification of additional CVD risk factors, enhances patient CVD awareness, increases physical activity, promotes a healthier diet, and improves wellbeing.

As the intervention evaluated in the trial consists of a bundle intervention including multiple interacting components, a process evaluation will be undertaken in parallel.

The investigators hypothesize that the bundle intervention will effectively reduce systolic and diastolic blood pressure and improve additional cardiometabolic and lifestyle-related factors. These factors are closely linked to the risk of future pregnancy complications and the development of vascular dysfunction.

STUDY DESIGN:

Population:

The investigators will recruit 760 first-time mothers in the early postpartum period with a preeclampsia diagnosis in their medical records, validated by research personnel. Women agreeing to participate in the trial will be invited to an in-person baseline visit (at home or in hospital) for baseline measurements and data collection. Participants will then be randomized in a 1:1 ratio to either the bundle intervention in addition to standard care, or standard care alone for the 9-month trial. Follow-up measurements and data collection will be conducted at 3 and 9 months for all participants.

Intervention:

A 9-month bundle intervention, consisting of evidence-based components aimed at enhancing cardiometabolic health, including targeted screening, self-monitoring, lifestyle modification, health education, motivational information, and support delivered via the trial-specific PEPP app (available for the intervention group only) and from health care study personnel. The PEPP-app's content partly builds on apps previously developed by our team members, focusing on physical activity, healthy dietary habits, and the integration of various behavior change techniques. It has been refined based on results from our feasibility study and patient representatives' input. The intervention starts with a Light phase and is followed by a more Intensive phase.

* Light phase (baseline-3 months): After randomization, the Light phase begins with an online visit with study healthcare personnel, for feedback from baseline measurements (e.g. targeted screening including blood pressure, blood glucose and blood lipids) as well as health education (e.g. preeclampsia and cardiovascular health). The app is then used for self-monitoring of blood pressure via a validated cellular-connected device, lifestyle modification (individual step count goals), health education (articles and podcasts), and support through chat and e-mail with study personnel. An online behavior modification group meeting with participants and study personnel will be held at about 1-2 months.
* Intensive phase (3-9 months): In addition to the features of the Light phase this phase includes an online visit with study healthcare personnel to provide feedback on 3-months screening results (targeted screening). It also introduces expanded features in the app on lifestyle modifications (individual goals for moderate-to-vigorous physical activity, a healthy-heart eating program to improve dietary quality), expanded health education, and additional self-monitoring of weight through a validated cellular-connected device. Online group meetings will be held during the intensive phase.

Control:

Standard care: Participants in the control group will receive standard postpartum care, in accordance with current clinical practices. According to Swedish guidelines. The control group will attend the trial visits for measurements at baseline and at 3 and 9-months follow-up.

ELIGIBILITY:
Inclusion Criteria

* First-time mothers postpartum
* Preeclampsia during first pregnancy
* Age ≥ 18 years
* Singleton live birth (infant still alive)
* Ability to understand and speak Swedish, English, Arabic, Somali, Dari, Persian, or Spanish
* Having a smartphone (Android or iOS)
* Ability to provide informed consent

Exclusion Criteria:

* Pre-pregnancy hypertension
* Diabetes mellitus type I or II
* Cardiovascular disease
* Kidney disease
* Systemic lupus erythematosus
* Antiphospholipid syndrome
* Previous or current eating disorders
* Ongoing new pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women who had preeclampsia during their first pregnancy
Enrollment: 760 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Change in systolic (sBP) blood pressure (mmHg) | From baseline to end of study at 9 months follow-up
  Change in systolic blood pressure (mmHg), recorded in single digits using a validated automatic blood pressure monitor.
Change in diastolic blood pressure (mmHg) | From baseline to end of study at 9 months follow-up
  Change in diastolic blood pressure (mmHg), recorded in single digits using a validated automatic blood pressure monitor.

SECONDARY OUTCOMES:
Change in postpartum weight (kilograms, kg) | From baseline to end of study at 9 months follow-up
  Change in postpartum body weight (kg), measured using a validated scale
Change in blood pressure (mmHg) stratified by early pregnancy BMI status | From baseline to end of study at 9 months follow-up
  Systolic and diastolic blood pressure (mmHg), recorded in single digits using a validated automatic blood pressure monitor. Early-pregnancy BMI will be calculated from weight (kg) and height (m) recorded in antenatal medical records by dividing the weight in kilograms by the square of the height in meters (kg/m²). Participants will be categorized into two subgroups based on BMI: <25 kg/m² and ≥25 kg/m². The outcome will be the mean change in blood pressure within each BMI subgroup.
Change in postpartum weight (kilograms, kg) by early pregnancy BMI status | From baseline to end of study at 9 months
  Change in postpartum body weight (kg), measured using a validated scale. Early-pregnancy BMI will be calculated from weight (kg) and height (m) recorded in antenatal medical records by dividing the weight in kilograms by the square of the height in meters (kg/m²). Participants will be categorized into two subgroups based on BMI: <25 kg/m² and ≥25 kg/m². The outcome will be change in postpartum body weight (kg) within each BMI subgroup.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Sandstrom, PhD, MD, Principal Investigator — Karolinska Institutet; Kari Johansson, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Stockholm County, Sweden